CLINICAL TRIAL: NCT00555243
Title: An Evaluation of Validated Laparoscopic Skills Simulators and the Impact on Operating Room Performance
Brief Title: Laparoscopic Simulator Training and Its Impact on Surgical Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Ochsner Health System (Other); University of Alabama at Birmingham (Other); The University of Texas Health Science Center, Houston (Other); Uniformed Services University of the Health Sciences (U.S. Federal Agency); Orlando Health, Inc. (Other); Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: UTSW IRB 042006-034
Record Dates: First submitted 2007-11-06; First posted 2007-11-08 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2007-11

CONDITIONS: Surgical Procedure, Unspecified; Surgical Simulation
Keywords: Laparoscopic Surgical Simulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Laparoscopic Simulation Education
  Interventions: Procedure: Laparoscopic Simulation training
- 2 (Placebo Comparator)
  Interventions: Procedure: Traditional Surgical Education

INTERVENTIONS:
Procedure: Laparoscopic Simulation training — five 30-minute faculty-directed sessions at the Laparoscopic Simulator Lab
  Other Names: Fundamentals of Laparoscopic Surgery
  Arms: 1
Procedure: Traditional Surgical Education — Traditional surgical teaching (no simulator)
  Arms: 2

SUMMARY:
The primary goal of this study is to answer whether validated laparoscopic simulators truly affect real time performance in the operating room among Gynecology residents.

DETAILED DESCRIPTION:
We have designed a randomized control trial to assess the impact of a laparoscopic simulator curriculum on operating room performance amongst gynecology residents. At the beginning of the study, each resident that chooses to participate will take a multiple choice pre-test assessing his or her background knowledge of laparoscopic surgical principles. Everyone will then listen to a series of lectures / video demonstrations teaching the fundamentals of laparoscopic surgery. The final part of the orientation is to have each resident perform 5 tasks on the laparoscopic simulators (peg transfer, endoloop, pattern cutting, intracorporeal suturing, and extracorporeal suturing) while being proctored by a faculty member who is timing the task and recording any errors made. Each resident will have 2 proctored performances (pre- and post) on the simulator and it will be set up as a typical OSCE-type exam. We chose to have them perform 2 repetitions as opposed to the usual 1 (like on the MCAT, SAT, or other high stake exam) to allow for potential unfamiliarity with the simulator equipment.

The residents will then perform a laparoscopic tubal ligation with a faculty member when they begin their Benign Gynecology rotation. Each resident will subsequently be randomized either traditional teaching (no simulator) or five 30-minute faculty-directed sessions at the Laparoscopic Simulator Lab. Those randomized to simulation training can practice and perform as many repetitions necessary on the simulator to achieve proficiency. Prior to completing the rotation, the residents will perform another laparoscopic tubal ligation with a faculty member blinded to whether they randomized to simulator training to re-assess their technical skills. The resident will have another proctored examination of simulator performance on the five tasks. Finally, a videotape review by independent observers will verify precision of the surgical evaluations at the conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

* All Ob/Gyn residents in post-graduate years 1-4 from ACGME accredited programs

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2005-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Whether laparoscopic simulators truly affect real time performance in the operating room among Gynecology residents | Over the course of one resident rotation (4-6 weeks)

SECONDARY OUTCOMES:
Determine if the level of improvement is inversely related to resident level of training. | Over the course of one resident rotation (4-6 weeks)
Calculate receiver operator curves to aid in the establishment of a "passing score" threshold on the validated laparoscopic simulators | Over the course of one resident rotation (4-6 weeks)
Establish whether psychomotor testing predicts surgical proficiency and helps identify those who may need more intensive training over the course of their education. | Over the course of one resident rotation (4-6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv B Gala, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (4):
- United States (4):
  - University of Alabama at Birmingham Department of Ob/Gyn, Birmingham, Alabama
  - Uniformed Services University of the Health Sciences, Washington D.C., District of Columbia
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas at Houston Department of Ob/Gyn, Houston, Texas

REFERENCES:
- [Derived] Gala R, Orejuela F, Gerten K, Lockrow E, Kilpatrick C, Chohan L, Green C, Vaught J, Goldberg A, Schaffer J. Effect of validated skills simulation on operating room performance in obstetrics and gynecology residents: a randomized controlled trial. Obstet Gynecol. 2013 Mar;121(3):578-584. doi: 10.1097/AOG.0b013e318283578b. PMID 23635621